CLINICAL TRIAL: NCT01991418
Title: Early Warning Study of Plasma Thioredoxin Reductase Activity in Non-small Cell Lung Cancers Received Surgery
Brief Title: Early Warning Study of Serum Thioredoixn Reductase Activity in Excised Non-small Cell Lung Cancers (EWSOTRILC)
Status: Completed | Type: Observational
Sponsor: Hunan Province Tumor Hospital (Other)
Responsible Party: Principal Investigator, Nong Yang, chief, Hunan Province Tumor Hospital
Other Study IDs: TR002; EWSOTRILC (Other: HunanPTH)
Record Dates: First submitted 2013-11-04; First posted 2013-11-25 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Non-small Cell Lung Cancer Stage I; Non-small Cell Lung Cancer Stage II; Non-small Cell Lung Cancer Stage IIIA
Keywords: non-small cell lung cancer; thioredoxin reductase; carcina embryonic antigen
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 3-4 ml whole blood was obtained and then centrifuged and stored at -20℃.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- early staged non-small cell lung cancer: patients diagnosed as early staged non-small cell lung cancer and received surgery in HunanPTH

SUMMARY:
In pre-clinical study, we found that serum thioredoxin reductase activity harbours huge difference after any kind of treatments, so we hypothesis that serum activity of thioredoxin reductase may be a warning markers in excised non-small lung cancers, serum activity of this enzyme may elevated before CT scan

DETAILED DESCRIPTION:
This is a cooperative research project in Thoracic Surgery Department and Medical Oncology department of Affiliated Cancer Hospital of xiangya School of Medicine Central South University, and the State Key Laboratory for Natural Medicine and Biomimetic Drugs Perking University. The primary objective is to measure the thioredoxin reductase activity in blood in staged(Ⅰ~ⅢA) non-small lung cancers, to study the warning relapse ability of thioredoxin reductase in blood. The secondary objective is to compare the warning relapse activity of blood thioredoxin reductase activity with carcinoembryonic antigen (CEA) in subjects who received surgery. Blood will be collected in subjects before surgery, 5 days after surgery, and every 3 months after surgery till 2 years, then every 6 months till 3 years, or collect blood till tumor relapse for the subjects at stage ⅠA and low risk ⅠB. Blood will be collected before surgery, 5 days after surgery, before adjuvant chemotherapy, after 2 circles of all adjuvant chemotherapy, then every 3 months after adjuvant chemotherapy till 2 years, and every 6 months till 3 years, or collect blood till tumor relapse for the subjects of high risk ⅠB~ⅢA, evaluation CT results every time collect blood samples.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically proven staged(Ⅰ~ⅢA) non-small cell lung cancer or CT scan shows resectable lung mass, fast pathology proved non-small cell lung cancer
* Receive surgery in Thoracic Oncology department Affiliated Cancer Hospital of xiangya School of Medicine Central South University without contraindication of surgery
* Tumor treatment naive（except for surgery for cervical cancer and cutaneous squamous cell carcinoma 5 years before）
* Signed informed consent to provide blood and tissue for study

Exclusion Criteria:

* Patients received antitumor treatment before
* Patients with contraindication of surgery or patients who need adjuvant chemotherapy with contraindication of chemotherapy
* Pregnant or breast feeding women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with resectable non-small lung cancer and received surgery in Affiliated Cancer Hospital of xiangya School of Medicine Central South University, HunanPTH
Sampling Method: Non-Probability Sample
Enrollment: 165 (Actual)
Dates: Start 2013-05; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Measure the thioredoxin reductase activity in blood | blood should be taken before and 3-5 days after surgery, then every 3 months till 2 years, then every 6 month till 3 years
  Measure the thioredoxin reductase activity in blood at the setting time point, before surgery, 3-5 days after surgery, after every 3 months after surgery till 2 years, then every 6 months till 3 years, or collect blood till tumor relapse in patients at stage ⅠA and low risk ⅠB. Blood will be taken before surgery, 3-5 days after surgery, before adjuvant chemotherapy, after two cycles of adjuvant chemotherapy, after every 3 months after adjuvant chemotherapy till 2 years, then every 6 months till 3 years, or collect blood till tumor relapse in patients at stage high risk ⅠB IIA IIB and IIIA.

SECONDARY OUTCOMES:
Measure carcina embryonic antigen(CEA) level in blood | blood should be taken before and 3-5 days after surgery, then every 3 months till 2 years, then every 6 month till 3 years
  Measure the carcina embryonic antigen(CEA) level in blood at the setting time point, before surgery, 3-5 days after surgery, after every 3 months after surgery till 2 years, then every 6 months till 3 years, or collect blood till tumor relapse in patients at stage ⅠA and low risk ⅠB. Blood will be taken before surgery, 3-5 days after surgery, before adjuvant chemotherapy, after two cycles of adjuvant chemotherapy, after every 3 months after adjuvant chemotherapy till 2 years, then every 6 months till 3 years, or collect blood till tumor relapse in patients at stage high risk ⅠB IIA IIB and IIIA.

CONTACTS AND LOCATIONS:
Overall Officials: Nong Yang, MD, Principal Investigator — Hunan Province Tumor Hospital
Locations (1):
- Hunan Provincal Tumor Hospital, Changsha, Hunan, China